CLINICAL TRIAL: NCT01535833
Title: Robotic Assisted Sacral Colpopexy : A Prospective Study Assessing Subjective and Objective Outcomes With Learning Curves in the Development of a New Pelvic Floor Robotics Program
Brief Title: Robotic Assisted Sacral Colpopexy : A Prospective Study Assessing Outcomes With Learning Curves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Shawn A Menefee, MD, Principal Investigator, Kaiser Permanente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP IRB 20111224
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: robotic sacral colpopexy; Learning curve; Pelvic Organ Prolapse; Robotic Surgery
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Robotic sacral colpopexy (Other): To assess subjects with stage 2 pelvic organ prolapse undergoing robotic sacral colpopex
  Interventions: Procedure: Device- Robotic sacral colpopexy

INTERVENTIONS:
Procedure: Device- Robotic sacral colpopexy — To assess robotic sacral colpopexy for female patients with stage 2 pelvic organ prolapse
  Other Names: Robotic Laparoscopic Sacral Colpopexy

SUMMARY:
The investigators scientific aims are to determine the benefits associated with the use of robotic assisted laparoscopic sacrocolpopexy surgery on women with prolapse, to define how the benefits impact the patient, physician and the institution, and to determine the complications associated with the use of the robot. This will be a prospective cohort following 100 patients for a 24 month period.

DETAILED DESCRIPTION:
The investigators scientific aims are to determine the benefits associated with the use of robotic assisted laparoscopic sacrocolpopexy surgery on women with prolapse, to define how the benefits impact the patient, physician and the institution, and to determine the complications associated with the use of the robot. This will be a prospective cohort following 100 patients for a 24 month period.

The investigators primary outcomes will be:

* Surgical time: Key portion of procedure will be assessed along with total time for completion
* Learning curve: Will be assessed using surgical times, VAS of camera skills, surgical skills involving tissue handling and movements and overall performance by surgeon, assistant and blind reviewer
* Length of hospitalization: measured by days in hopsital

The investigators secondary outcomes will be:

* Pre-operative and postoperative Pelvic Organ Prolapse-Quantification (POP-Q) at 6 week, 6, 12, and 24 months.
* Pelvic Floor Distress Inventory-Short Form 20 Questionnaire (PFDI-20)
* Mesh erosion,
* Estimated blood loss,
* Complications (bowel or bladder injury) and,
* Wound infection,
* Patient Global Impressions of Improvement
* Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Females only
* Undergoing robotic assisted laparoscopic sacrocolpopexy with or without other procedures for pelvic organ prolapse
* Willing to return for follow-up visits
* Written informed consent obtained from each subject

Exclusion Criteria:

* Decline to participate
* Pregnant or contemplating future pregnancy (within a year)
* Unable to participate in the informed consent process

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Learning curve of robotic sacral colpopexy | 24 months
  To assess learning curve during implementation of a new pelvic floor robotic program which will assess surgical time (total and specific essential portions), simulator training and surgeon, observational surgeon skills by surgeon, assistant and blinded assessor

SECONDARY OUTCOMES:
Subjective outcomes for robotic sacral colpopexy | Two years
  Subjective outcomes for robotic sacral colpopexy for prolapse and incontinence symptoms and sexual function using validated measures (PFDI-20), (PISQ-12)
Adverse events for robotic sacral colpopexy | Two years
  Adverse events for robotic sacral colpopexy including estimated blood loss, GU and GI injury, wound infection and mesh erosion
Objective outcomes measures associated with robotic sacral colpopexy | 24 months
  To assess prolapse outcomes using POP-Q assessment of postoperative support at 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Brown, Study Director — Southern California Kaiser permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Downey, Los Angeles, California
  - Kaiser Permanente San Diego, San Diego, California